CLINICAL TRIAL: NCT06220578
Title: Analysis of Topographic Corneal Parameters in a Large Cohort of Corneal Refractive Surgery Candidates
Brief Title: Analysis of Topographic Corneal Parameters
Status: Completed | Type: Observational
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahemd Abdelghany, Associate professor, Minia University
Other Study IDs: 592/2023
Record Dates: First submitted 2024-01-12; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Cornea
MeSH Terms: conditions — Corneal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- candidates seeking corneal refractive surgery: Persons from both sexes between 18 and 45 years seeking corneal refractive surgery
  Interventions: Device: Oculus pentacam HR

INTERVENTIONS:
Device: Oculus pentacam HR — Examination of corneal parameters by pentacam

SUMMARY:
The Pentacam HR system (OCULUS) has been suggested to be one of the most sensitive instruments for corneal examination before corneal refractive surgery

DETAILED DESCRIPTION:
Retrospective non randomized study Analysis of different corneal paremeters obtained by Pentacam for corneal refractive surgery candidates during last 3 years from both sexes between 18 and 45 years K1 - K2 - K max - Pachymetry apex - Pachymetry thinnest - Distance between apex and thinnest - Back elevation - Topography shape - Keratoconus (If present)

ELIGIBILITY:
Inclusion Criteria:

* Persons from both sexes between 18 and 45 years seeking corneal refractive surgery

Exclusion Criteria:

* Previous intraocular surgery
* Previous corneal surgery
* Corneal opacity

Ages: 18 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: patients examined in Roaa LASIK center from both sexes between 18-45 years seeking corneal refractive surgery
Sampling Method: Non-Probability Sample
Enrollment: 2694 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
corneal curvature | 7 months
  radii of curvature in diopters
corneal pachymetry | 7 months
  measured in microns

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdelghany, professor, Principal Investigator — Minia University
Locations (1):
- Faculty of Medicine, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No
not plan to share